CLINICAL TRIAL: NCT05652413
Title: Enhancing Recruitment and Engagement of African American Older Adults With Osteoarthritis Pain in a Behavioral Pain Management and Physical Activity Intervention
Brief Title: Engaging African American Older Adults With Arthritis in a Physical Activity Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00108300
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Osteoarthritis, Knee; Osteoarthritis, Hip
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adapted-Engage-PA (Experimental): Participants will receive two sessions, lasting 60 minutes each, of behavioral intervention strategies to increase daily walking routines and prevent pain flares.
  Interventions: Behavioral: Adapted-Engage-PA

INTERVENTIONS:
Behavioral: Adapted-Engage-PA — Enhanced motivation strategies for increasing walking using personal values assessment and value-guided goal setting, adapted from Acceptance and Commitment therapy. Strategic activity pacing to increase stamina and reduce pain flares when walking, using the Activity Rest Cycle, from Pain Coping Skills Training. Culturally sensitive elements for older adults who identify as African American such as linking motivation to spirituality, family, community, and other personally-meaningful values.

SUMMARY:
Physical activity like walking is one important way to reduce pain and improve wellbeing for older adults with knee and hip arthritis, but most older adults and particularly those who identify as African American struggle to walk regularly. Many African Americans with arthritis have worse outcomes (like worse pain, worse overall health) than other racial and ethnic groups for many reasons including racist policies and ideas that make getting good health care more difficult. It is therefore most important to identify ways to help older adults who identify as African American improve their arthritis pain and improve their daily steps. The current study is designed to learn about older African American's preferences for a brief behavioral intervention to increase daily steps and reduce pain, and to learn about the barriers (things that make walking harder) and facilitators (things that make walking easier) for walking that they experience. Interviews with both patients and healthcare providers will provide important information that will be used to adapt an existing behavioral intervention designed to help patients increase their daily steps and reduce their arthritis pain. The final adapted intervention will be tested in a small clinical trial with older adults who identify as African American to see if it can reduce pain and increase walking over time.

DETAILED DESCRIPTION:
Osteoarthritis is one of the most common risk factors for disability for African American older adults. Older adults who identify as African American experience more severe arthritis, higher pain levels, more pain related interference, more health problems that occur alongside arthritis, and have greater problems accessing appropriate and timely care for arthritis than other racial and ethnic groups. Physical activity can help improve pain and is safe even for older adults, but few older adults walk regularly due to pain, psychological distress, and other environmental barriers for walking. Specific strategies targeted to support older African Americans in walking more are needed. A previously tested behavioral intervention called Engage-PA has shown promise for supporting older adults with arthritis in the knee and/or hip. Yet little is know about how promising this intervention is for older African Americans, nor the specific barriers and facilitators for walking more for this population. Some specific components of Engage-PA may be particularly culturally-relevant for older African Americans, such as the use of personal values, or a detailed discussion of personally-identified meaning and purpose linked to daily walking routines. Older African Americans with arthritis and primary care providers treating arthritis at Duke Health have provided interview data to assist researchers in adapting Engage-PA to be more culturally sensitive. Adapted-Engage-PA will be tested with older African Americans who have knee and/or hip pain from osteoarthritis in a small feasibility and acceptability trial.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 or older
2. English speaking
3. identify as Black/African American
4. diagnosis of osteoarthritis in knee or hip
5. able to ambulate even if assisted with walker or cane
6. endorse worst pain and pain interference as ≥ 3 out of 10 within the last week

Exclusion Criteria:

1. hearing or visual impairment that would prevent ability to participate in sessions or use participant worksheets, even with use of adaptive supports/devices
2. planned surgery during study duration that would limit mobility (e.g., due to recommended rehabilitation or recovery period) for more than 3 weeks
3. current enrollment in cardiac rehabilitation
4. myocardial infarction in the past 3 months
5. major surgery requiring limited movement or mobility for recovery within the past 3 months
6. presence of a serious psychiatric condition (e.g., schizophrenia, suicidal intent) that would contraindicate safe study participation
7. Medical provider indicating that exercise (even walking) should only be medically supervised
8. fall or falls within the last 3 months that led to immediate medical treatment/hospitalization
9. reported or suspected moderate or severe cognitive impairment
10. brain tumor/cancer metastases to the brain
11. no other conditions that would preclude safe participation (e.g., unmanaged heart conditions, neurodegenerative condition, unmanaged diabetes, severe respiratory disease), as screened the Physical Activity Readiness Questionnaire (PAR-Q+ 2020, a measure widely utilized by the U.S. National Academy of Sports Medicine and the Public Health Agency of Canada). Answers to the PARQ+2020 may result in review by patient physicians for safety prior to enrollment.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Number of enrolled participants | 6 months
  Did the study reach full anticipated accrual?
Number of participants who completed the entire program | 8 weeks
  Participants who complete all assessments and required study sessions
Percentage of participants who were mostly or very satisfied with the intervention | Post-treatment (8 weeks)
  Client Satisfaction Questionnaire asks 8 questions related to patient satisfaction on a Likert Scale of 1= very satisfied to 7 = very dissatisfied. There is one item assessing overall satisfaction with the intervention, and the percentage of participants responding to this item with "mostly" or "very" satisfied is reported below.

SECONDARY OUTCOMES:
Arthritis Pain (AIMS 2 Symptom Subscale) | Baseline, post-treatment (8 weeks)
  The Arthritis Impact Measurement Scale (AIMS 2) measures arthritis pain related disability across areas of living both with a total score and on several subscales (i.e., pain severity, physical functioning/pain- related disability, psychological distress), where 1 indicates very good functioning, and 5 indicates very poor functioning. Symptom subscale includes items assessing pain severity, stiffness, and physical discomfort. Range is 5 to 25 where higher scores indicate worse functioning.
Arthritis-related Physical Functioning (AIMS 2 Physical Functioning Subscale) | Baseline, post-treatment (8 weeks)
  The Arthritis Impact Measurement Scale (AIMS 2) measures arthritis pain related disability across areas of living on several subscales (i.e., pain severity, physical functioning/pain-related disability, psychological distress), where 1 indicates very good functioning, and 5 indicates very poor functioning. Physical functioning subscale includes items assessing mobility level, walking and bending, self-care and household tasks. Range is 5-25 where higher scores indicate worse functioning.
Psychological Distress (AIMS 2 Affect Subscale) | Baseline, post-treatment (8 weeks)
  The Arthritis Impact Measurement Scale (AIMS 2) measures arthritis pain related disability across areas of living on several subscales (i.e., pain severity, physical functioning/pain-related disability, psychological distress), where 1 indicates very good functioning, and 5 indicates very poor functioning. Psychological distress subscale includes items assessing mood and anxiety/tension. Range is 5-25 where higher scores indicate worse functioning.
Step Count | Baseline, post-treatment (8 weeks)
  Daily step counts as reported to study staff, after participants recorded them from wearable fitness trackers at end of day. Each assessment period consisted of 7 continuous days of wear. Summed totals of steps in the 7 day period were calculated, and then means calculated between groups of these summed step counts for the 7 day assessment period.
Rapid Assessment of Physical Activity | Baseline, post-treatment (8 weeks)
  The RAPA is a self-reported measure that assesses participants engagement in a variety of activities, such as light movement, moderate activity, vigorous activity, and other activities such as strength-training or yoga. Scores range from 0 - 7, where higher scores indicate greater involvement in physical activity overall.
Psychological Flexibility | Baseline, post-treatment (8 weeks)
  The Acceptance and Action Questionnaire-II asks about psychological flexibility, defined as how often thoughts, feelings and body sensations get in the way of living a fulfilling life. Responses are on a 1 to 7 Likert scale with 1 indicating that these issues never get in the way, and 7 indicating that these issues always get in the way. Range is 7 - 49, with lower scores indicating better outcomes.
  Title: Psychological Flexibility The Acceptance and Action Questionnaire-II asks about psychological flexibility, defined as how often thoughts, feelings and body sensations get in the way of living a fulfilling life. Responses are on a 1 to 7 Likert scale with 1 indicating that these issues never get in the way, and 7 indicating that these issues always get in the way. Range is 7 - 49, with lower scores indicating better outcomes.
Valued Living - Health Domain | Baseline, post-treatment (8 weeks)
  The Bulls-Eye Values measure assesses how successfully participants are at living in line with 4 domains of personal values (relationships, leisure, health, and work) on a visual dart-board scale with 1 indicating perfect success, and 14 indicates being unsuccessful. Range for each domain is 1 - 14 with lower as better outcome.
Valued Living - Leisure Domain | Baseline, post-treatment (8 weeks)
  The Bulls-Eye Values measure assesses how successfully participants are at living in line with 4 domains of personal values (relationships, leisure, health, and work) on a visual dart-board scale with 1 indicating perfect success, and 14 indicates being unsuccessful. Range for each domain is 1 - 14 with lower as better outcome.
Valued Living -Relationship Domain | Baseline, post-treatment (8 weeks)
  The Bulls-Eye Values measure assesses how successfully participants are at living in line with 4 domains of personal values (relationships, leisure, health, and work) on a visual dart-board scale with 1 indicating perfect success, and 14 indicates being unsuccessful. Range for each domain is 1 - 14 with lower as better outcome.
Valued Living -Work/Community Domain | Baseline, post-treatment (8 weeks)
  The Bulls-Eye Values measure assesses how successfully participants are at living in line with 4 domains of personal values (relationships, leisure, health, and work) on a visual dart-board scale with 1 indicating perfect success, and 14 indicates being unsuccessful. Range for each domain is 1 - 14 with lower as better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Plumb Vilardaga, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No